CLINICAL TRIAL: NCT02904824
Title: Injection Laryngoplasty Using Autologous Fat Enriched With Adipose Derived Regenerative Stem Cells (ADRC) vs Centrifuged Autologous Fat (CAF), for the Functional Reconstruction of the Glottal Gap After Unilateral Vocal Cord Paralysis
Brief Title: Injection Laryngoplasty Using Autologous Fat Enriched With Adipose Derived Regenerative Stem Cells (ADRC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIBHGM-ECNC007-2010
Record Dates: First submitted 2016-07-20; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Vocal Cord Paralysis, Unilateral
Keywords: adipose tissue; adult stem cells; vocal cord paralysis
MeSH Terms: conditions — Vocal Cord Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ADRC, adipose derived regenerative cells (Experimental): Biological: Stem cells from autologous adipose tissue in which autologous tissue is enriched or in suspension to fill the paralyzed vocal cord. The aim is to induce the overexpression and production of microvessels at local level. Route of administration: injection into the thickness of a paralyzed vocal cord.
  Interventions: Biological: adipose derived regenerative cells
- CAF, centrifuged autologous fat (Active Comparator): Biological: Autologous fat tissue processed by centrifugation. Route of administration: Injection inside a paralyzed vocal cord.
  Interventions: Biological: centrifuged autologous fat

INTERVENTIONS:
Biological: adipose derived regenerative cells — Stem cells from autologous adipose tissue in which autologous tissue is enriched or in suspension to fill the paralyzed vocal cord. The aim is to induce the overexpression and production of microvessels at local level. Route of administration: injection into the thickness of a paralyzed vocal cord.
  Arms: ADRC, adipose derived regenerative cells
Biological: centrifuged autologous fat — centrifuged adipose tissue which is autologous tissue is used to fill the paralyzed vocal cord. The aim is to increase the volume of the vocal fold, to reduce the glottal gap.This effect is temporary. Route of administration: injection into the thickness of a paralyzed vocal cord.
  Arms: CAF, centrifuged autologous fat

SUMMARY:
This is the first Development Safety Update Report prepared for Phase I-IIA Clinical Trial- FIBHGM-ECNC007-2010 (PHASE I / IIA CLINICAL TRIAL, UNICENTRIC, RANDOMIZED, CONTROLLED, TWO PARALLEL-GROUPS, TO EVALUATE THE SAFETY OF A NEW THERAPY WITH STEM CELLS DERIVED FROM ADIPOSE TISSUE FOR GLOTTAL GAP(GG) IN THE UNILATERAL PARALYSIS OF THE VOCAL CORD(VC) ) in the International Conference on Harmonization (ICH). Patients are randomized to receive one of the following therapeutic strategies:

Group A: Autologous Fat processed by centrifugation to fill a paralyzed vocal cord. Group B: Autologous Fat enriched with stem cells from adipose tissue to treat vocal cord paralysis.

Active control: Autologous fat tissue processed by centrifugation. Route of administration: Injection into a paralyzed vocal cord.

Experimental drug: Stem cells from autologous adipose tissue in which autologous tissue is enriched or in suspension to fill the paralyzed vocal cord. The aim is to induce the overexpression and production of microvessels at local level. Route of administration: injection into the thickness of a paralyzed vocal cord.

DETAILED DESCRIPTION:
This is the first Development Safety Update Report prepared for Phase I-IIA Clinical Trial- FIBHGM-ECNC007-2010 (PHASE I / IIA CLINICAL TRIAL, UNICENTRIC, RANDOMIZED, CONTROLLED, TWO PARALLEL-GROUPS, TO EVALUATE THE SAFETY OF A NEW THERAPY WITH STEM CELLS DERIVED FROM ADIPOSE TISSUE FOR GLOTTAL GAP IN THE UNILATERAL PARALYSIS OF THE VOCAL CORD in the International Conference on Harmonization (ICH) E2F format. This trial contains relevant safety information from the reporting interval of 08 July 2012 to 30 Sep 2014 This phase I / IIA clinical trial has been conducted to evaluate the safety of ADRCs. This new therapy is performed to induce the overexpression and production of microvessels in the paralyzed vocal cord, to permanently increase its volume and thus facilitate the GG closure. In paralysis of VC an increase of glottal gap occurs leading to dysphonia and aspiration of food, foreign bodies...

The creation of these new blood vessels, through the action of stem cells derived from adipose tissue, may produce a greater volume of the paralyzed vocal cord allowing GG closure more easily.

Patients included in this clinical trial require treatment for unilateral vocal cord paralysis. It has been considered regarding the authorised protocol that a glottal GAP requires intracordal injection to increase its volume when the glottal closure·during phonation is insufficient or there is lack of compensation to the contralateral vocal cord.

Patients are randomized to receive one of the following therapeutic strategies:

Group A: Autologous Fat processed by centrifugation to fill a paralyzed vocal cord, using the same.

Group B: Autologous Fat enriched with stem cells from adipose tissue to treat vocal cord paralysis.

Active control: Autologous fat tissue processed by centrifugation. Route of administration: Injection inside a paralyzed vocal cord.

Experimental drug: Stem cells from autologous adipose tissue in which autologous tissue is enriched or in suspension to fill the paralyzed vocal cord. The aim is to induce the overexpression and production of microvessels at local level. Route of administration: injection into the thickness of a paralyzed vocal cord.

In patients assigned to ADRC group therapy, two surgical interventions are performed on the same day, once randomized, at visit 0 according to the protocol. For the group assigned to the control (autologous adipose tissue), the therapy is performed in a single surgical intervention, once randomized, at visit 0 according to protocol.

The patients who are included will be followed for six months from the implant.

ELIGIBILITY:
Inclusion Criteria:

* VC paralysis in paramedian position.
* Patients without previous compensation of the healthy contralateral VF.
* Males and females 18-years old or older.
* Women presenting the possibility of being pregnant must present a negative test of current pregnancy before the inclusion in the clinical trial (it must be certified at the minus 2 medical visit). It can be done by a blood test or a urinary test.
* The paralyzed VC should not be affected by granulomas, tumors o macroscopic objectable lesions by conventional laryngoscopy.
* The clinical situation of the patient must be ASA I or II following the parameters of the American Society of Anesthesiologists.
* There should not be any circumstance that could not afford the patient to follow the procedures of the clinical trial at least 6 months from the operation day.
* The patient must sign and confirm a specific informed acceptance to participate in the trial

Exclusion Criteria:

* Patients affected by kidney insufficiency, presenting a seric creatinine higher than 2.5 mg/dl.
* Medical history of allergy to proteins, or other allergies that could lead to a safety problem if the patient joins the present clinical trial.
* Acute infectious disease at the moment of enrollment.
* Chronic infectious disease affecting directly or indirectly the anatomical area that is going to be operated (it includes tuberculosis, brucellosis, chronic candidiasis and cutaneous chronic ulcers).
* Pregnancy or lactating patient.
* Patient needing a surgery in the anatomical area that is going to be operated on for a different reason at the moment of inclusion in the study, or patients in which it is suspected to perform surgeries in the mentioned anatomical area 24 weeks after the implant.
* Alcohol abuse or drugs abuse 6 months before the inclusion.
* Latent or active HIV infection or viral hepatitis.
* Patient suffered a major surgery or a major trauma 28 days before enrollment.
* Patients treated with immune-modulators (including therapy with systemic stem cells) 6 months before the inclusion in the study.
* Lung or heart disease that is unstable of presents a gravity that suggests to exclude the enrollment in the study.
* Life expectancy inferior to one year, in relation to comorbidities presenting in the moment of the clinical evaluation.
* Patients presenting deep venous thrombosis or lung thromboembolism, or patients who presented these diseases 6 months before the inclusion in the study.
* Patient presenting acquired or congenital immunodeficiencies.
* Patients presenting hemorrhagic diseases with INR>2,0, without anticoagulant treatment.
* Patients with any medical or psychiatric disorder that under the point of view of the researchers justifies the exclusion in the trial, because follow-up could be interrupted, because enrolment could be a risk for the patient or because it could be a risk for the global evaluation of the clinical trial.
* Patients enrolled currently in other clinical trials, or patients that participated in clinical trial 30 days before the inclusion in this study, if the previous one could not interfere in the participation or in the evaluation of the objectives of the present study.
* Patient who does not wish or cannot follow the procedures indicated in the clinical trial.
* Patients treated with platelet anti-aggregates or non-steroid anti-inflammatories 15 days before the surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-07; Primary Completion 2014-09 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | up to 6 months
  Adipose derived stem cells injected into the vocal cords are evaluated in order to study the incidence of possible adverse events: Glottal oedema, laryngospasm, granuloma at the vocal cord, anaphylactic shock, induced tumorigenesis are undesirable adverse events.

SECONDARY OUTCOMES:
Assessment of vocal cord volume and gap closure by direct laryngoscopy and Biometphone device to study vocal cord parameters | up to 6 months
  Direct laryngoscope will evaluate the volume of the paralyzed one and measure the GG. The description of the GG conditions observed in patients before and after the treatment from laryngoscopy inspections prior and 180 days after surgery may show incomplete coaptations of the GG presenting a partial closure pattern or total coaptation.
  Biomet phone is a device that measures biomechanical characterization of voice. Accurate spectral domain techniques allow the estimation of a set of biomechanical parameters associated to a 2-mass model of the VF from the glottal source spectral density.
  The modification in voice quality can be expressed numerically using likelihood estimations. In evaluating the improvement in voice quality, the proposed methodology is based on the use of the Log Likelihood Improvement Ratios (LLIR), a metrics founded on alternative hypothesis testing speech evidence matching.

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Lasso, MD, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañón
Locations (1):
- Jose M Lasso, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu M, Zhou Z, Chen Y, Schreiber R, Ransom JT, Fraser JK, Hedrick MH, Pinkernell K, Kuo HC. Supplementation of fat grafts with adipose-derived regenerative cells improves long-term graft retention. Ann Plast Surg. 2010 Feb;64(2):222-8. doi: 10.1097/SAP.0b013e31819ae05c. PMID 20098110
- [Background] Perez-Cano R, Vranckx JJ, Lasso JM, Calabrese C, Merck B, Milstein AM, Sassoon E, Delay E, Weiler-Mithoff EM. Prospective trial of adipose-derived regenerative cell (ADRC)-enriched fat grafting for partial mastectomy defects: the RESTORE-2 trial. Eur J Surg Oncol. 2012 May;38(5):382-9. doi: 10.1016/j.ejso.2012.02.178. Epub 2012 Mar 15. PMID 22425137
- [Background] Rosen CA, Lee AS, Osborne J, Zullo T, Murry T. Development and validation of the voice handicap index-10. Laryngoscope. 2004 Sep;114(9):1549-56. doi: 10.1097/00005537-200409000-00009. PMID 15475780
- [Background] Gómez P, Fernández R, Rodellar V, Nieto V, Álvarez A, Mazaira LM, Martínez R., Godino JI. Glottal Source Biometrical Signature for Voice Pathology Detection, Speech Communication; 51 2009, pp 759-781.
- [Background] Cantarella G, Mazzola RF, Domenichini E, Arnone F, Maraschi B. Vocal fold augmentation by autologous fat injection with lipostructure procedure. Otolaryngol Head Neck Surg. 2005 Feb;132(2):239-43. doi: 10.1016/j.otohns.2004.09.022. PMID 15692533
- [Derived] Lasso JM, Poletti D, Scola B, Gomez-Vilda P, Garcia-Martin AI, Fernandez-Santos ME. Injection Laryngoplasty Using Autologous Fat Enriched with Adipose-Derived Regenerative Stem Cells: A Safe Therapeutic Option for the Functional Reconstruction of the Glottal Gap after Unilateral Vocal Fold Paralysis. Stem Cells Int. 2018 Apr 15;2018:8917913. doi: 10.1155/2018/8917913. eCollection 2018. PMID 29760737
- Available data/document: Clinical Study Report — http://www.dynasolutions.com — CRO data base